CLINICAL TRIAL: NCT07206160
Title: Effect of Dapagliflozin on Interleukin 10 Compared to High Density Lipoprotein As a Prognosis in Septic Patients
Brief Title: Effect of Dapagliflozin on Interleukin 10 in Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mostafa Ragab Lokai Shahat, Assistant lecturer of Anesthesia and Intensive Care, Minia University
Other Study IDs: Dapagliflozin in sepsis
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group (D) will receive dapagliflozin 10mg tablet and Group (C) will receive vitastress tablet

SUMMARY:
The goal of this observational study is to learn about the long-term effects of dapagliflozin as anti-inflammatory agents to improve organ dysfunction and decrease mortality on patients of both genders ageing 18 years or above with sepsis.

1ry Outcome: The anti-inflammatory effect of dapagliflozin in patients with sepsis evaluated by: Effect on inflammatory markers (IL-10).

2ry Outcomes:

1. Severity of sepsis evaluated by the SOFA score.
2. Prognostic value of HDL compared to IL-10 for multi organ failure and death in septic patients and their correlation to the severity of sepsis.
3. ICU mortality &hospital length stay.

DETAILED DESCRIPTION:
64 Patients fulfilling the criteria for sepsis admitted to ICU will be allocated into 2 groups (32 patients in each group):

* Dapagliflozin group: Patients will receive dapagliflozin at a dosage of 10mg mixed with 10ml water at the time of admission for 7 days (or until ICU discharge, whichever comes first).
* Placebo group: Patients will receive vitastress tab .

The solutions of the study medications will be prepared by a hospital pharmacist and the medication will be administrated through the nasogastric tube in patients with disorder of consciousness or swallowing deficit.

Dapagliflozin will be stopped if the patients enter in more than one episode of severe hypoglycemia (≤50mg/dL) or occurrence of euglycemic diabetic ketoacidosis, defined by high anion gap metabolic acidosis and ketone bodies in the urine. Also the drug will be withheld if idiosyncratic drug reactions, such as DRESS syndrome (drug rash with eosinophilia and systemic symptoms) or allergic reaction to dapagliflozin has been occurred and if there is any need for absolute fasting and/or inability to access the enteral route for the drug.

ELIGIBILITY:
Inclusion Criteria:

* 64 adult patients of both sex, over the age of 18 years who were admitted to the ICU with sepsis and those who developed sepsis in the ICU.

Exclusion Criteria:

- 1. Patient's refusal, pregnant and lactating patients. 2. Known allergy or intolerance to dapagliflozin. 3. Unable to receive enteral medication& patients with chronic liver disease. 4. Shock 5. Patients with malabsorption disorders & or receipt of total parenteral nutrition and on treatment with statins.

6. Patients with a history of familial hyperlipidemia. 7. End-stage renal disease (ESRD) on regular dialysis. 8. Type 1 diabetes.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 64 adult patients of both sex, over the age of 18 years who diagnosed with sepsis which meet the criteria: Suspicious/ known infection/ Increase of ≥ 2 SOFA score with elevated white blood cells and C reactive protein and inflammatory markers.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
the anti-inflammatory effect of dapagliflzin | 7 days
  Effect on inflammatory markers (IL-10).
The anti-inflammatory effect of dapagliflozin in patients with sepsis | baseline
  Effect of dapagliflozin in sepsis evaluated by: Effect on inflammatory markers (IL-10).

REFERENCES:
- [Background] Dellinger RP, Carlet JM, Masur H, Gerlach H, Calandra T, Cohen J, Gea-Banacloche J, Keh D, Marshall JC, Parker MM, Ramsay G, Zimmerman JL, Vincent JL, Levy MM; Surviving Sepsis Campaign Management Guidelines Committee. Surviving Sepsis Campaign guidelines for management of severe sepsis and septic shock. Crit Care Med. 2004 Mar;32(3):858-73. doi: 10.1097/01.ccm.0000117317.18092.e4. PMID 15090974
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- See also: Related Info — https://www.sccm.org/clinical-resources/guidelines/guidelines/surviving-sepsis-guidelines-2021